CLINICAL TRIAL: NCT01210261
Title: New Versus Existing Auto-titrating CPAP Device to Treat Obstructive Sleep Apnea in Adults: Randomised Non-inferiority Double Blinded Trial.
Brief Title: New Versus Existing Auto-titrating CPAP Device to Treat Obstructive Sleep Apnea in Adults
Acronym: APAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Compumedics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPAP001; 10244A (Other: Southern Health, Monash Medical Centre, Research Project No.)
Record Dates: First submitted 2010-09-23; First posted 2010-09-28 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: OSA; CPAP; APAP; SPAP; Obstructive Sleep Apnea; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autoset S8 (Active Comparator): Single night auto-titrating CPAP treatment using the reference device (Resmed Autoset S8) with polysomnographic monitoring
  Interventions: Device: Resmed Autoset S8 - Auto-titrating CPAP
- Somnilink SPAP (Experimental): Single night auto-titrating CPAP treatment using the test device with polysomnographic monitoring
  Interventions: Device: Compumedics Somnilink SPAP - Auto-titrating CPAP

INTERVENTIONS:
Device: Compumedics Somnilink SPAP - Auto-titrating CPAP — Subjects will undergo the auto-titrating CPAP treatments in the Monash Sleep Centre with the test and reference devices during two nights in random order. There will be an interval of at least seven days between the two treatments to eliminate the carryover effect.
  Full polysomnographic (PSG) recording will be conducted during both treatment nights. The recorded physiological signals during PSG will include signals identical to those used during the baseline diagnostic PSG. The patients fill KSS questionnaire immediately after the PSG study.
  All PSG recordings (both treatment studies and the baseline diagnostic study) will be scored according to the AASM rules by the same sleep technician blinded to the presence and type of auto-titrating CPAP treatment.
  Other Names: Somnilink SPAP
  Arms: Somnilink SPAP
Device: Resmed Autoset S8 - Auto-titrating CPAP — Subjects will undergo the auto-titrating CPAP treatments in the Monash Sleep Centre with the test and reference devices during two nights in random order. There will be an interval of at least seven days between the two treatments to eliminate the carry-over effect.
  Full polysomnographic (PSG) recording will be conducted during both treatment nights. The recorded physiological signals during PSG will include signals identical to those used during the baseline diagnostic PSG. The patients fill KSS questionnaire immediately after the PSG study.
  All PSG recordings (both treatment studies and the baseline diagnostic study) will be scored according to the AASM rules by the same sleep technician blinded to the presence and type of auto-titrating CPAP treatment.
  Other Names: Autoset S8
  Arms: Autoset S8

SUMMARY:
Obstructive sleep apnea (OSA) is a condition of disordered breathing characterised by intermittent partial and/or complete upper airway obstruction during sleep. The participants, naive to nasal continuous positive airway pressure (CPAP), recently diagnosed with OSA, will undergo two automatic CPAP titration studies with collection of polysomnographic (PSG) data. The data will be analysed to assess effectiveness of Compumedics auto-CPAP device in the normalisation of sleep disordered breathing in OSA patients, with respect to another auto-CPAP device.

DETAILED DESCRIPTION:
Auto-titrating CPAP (APAP) using algorithms based on detection of flow limitation and snoring have been developed. Auto-titration devices adjust nasal pressure to the minimum pressure needed to maintain airway patency at any point in time and can accommodate a range of background states that affect airway collapsibility and hence CPAP pressure requirement including sedation, alcohol, airway inflammation, body position and sleep state.

Compumedics Limited has developed an APAP device (Somnilink SPAP based on the new algorithm technology of characterising breaths and determination of inspiratory flow limitation. The objectives of this new technology are to enable accurate detection of inspiratory intervals for irregular breathing patterns that are likely to occur during REM sleep, sleep onset and wakefulness as well as to provide correct characterisation of inspiratory flow limitation. These features could translate in delivery of superior treatment because of improved sensitivity and specificity of respiratory event detection and earlier pressure response to inspiratory flow limitation. Demonstration of superiority of the Somnilink SPAP device relative to existing APAP treatment devices will be subject of future clinical trials (beyond the scope of this protocol). An early clinical trial of a pre-production version of Somnilink SPAP with the pressure control algorithm identical to the production version established non-inferiority for AHI relative to a reference APAP (Resmed Autoset Spirit) with the differential AHI estimate of -0.91 [-2.80; 0.91] (Mean [95%CI]). The Somnilink SPAP device is now available as a production version (CE and TGA approved) and the purpose of the current study is to establish its non-inferiority compared to an existing APAP device (Resmed Autoset S8).

The treatment will be administered on the two nights of polysomnographic studies (PSG) by means of continuous air pressure delivery under the variable pressure levels determined by the APAP device to maintain the upper airway patency.

The population of adult patients newly diagnosed with OSA after undergoing a diagnostic PSG study in the sleep laboratory with no previous CPAP treatment experience and complying with the eligibility criteria (as outlined below) will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18.
* Ability to give informed consent.
* OSA diagnosis and referral for clinical CPAP implementation at the Monash Sleep Centre within 3 months of recruitment.

Exclusion Criteria:

* Inability to give informed consent.
* Significant central sleep apnea (AHI for central events >= 5).
* Congestive heart failure.
* Co-existing obesity related hypoventilation.
* Nasal obstruction, mouth breathing or other anatomical or physiological conditions making CPAP therapy inappropriate.
* History of prior CPAP treatment.
* Previous reaction to skin preparation, tapes and electrode gels used at PSG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) difference between test and reference APAP treatment | Up to 8 weeks after study completion
  AHI is the number of apnea and hypopnea events per hour of sleep

SECONDARY OUTCOMES:
AHI difference between test treatment and baseline | Up to 8 weeks after study completion
  AHI is the number of apnea and hypopnea events per hour of sleep.
  This endpoint is introduced to further demonstrate effectiveness of the test treatment in addition to the body of knowledge deduced from historical evidence for the reference treatment and selection conditions of the margin of non-inferiority
Arousal Index (AI) differences between the test and reference APAP treatments and between the test treatment and baseline | Up to 8 weeks after study completion
  AI is the number of occurrences of arousal events per hour of sleep.
  AI differences will be tested between test and control as non-inferiority, and between test and baseline as superiority.
Respiratory Disturbance Index (RDI) differences between the test and reference APAP treatments and between the test treatment and baseline | Up to 8 weeks after study completion
  RDI is the number of respiratory events (apneas and hypopneas) and respiratory event related arousals (RERA) [39] per hour of sleep.
  RDI will be tested between test and control as non-inferiority, and between test and baseline as superiority.
Sleep Efficiency (SE) differences between the test and reference APAP treatments and between the test treatment and baseline | Up to 8 weeks after study completion
  SE is defined as the ratio of sleep time to the time in bed.
  SE will be tested between test and control as non-inferiority, and between test and baseline as superiority.
Oxygen desaturation index (DI) differences between the test and reference APAP treatments and between the test treatment and baseline | Up to 8 weeks after study completion
  DI is defined as the number of oxygen desaturations >= 3% per hour of sleep.
  DI will be tested between test and control as non-inferiority, and between test and baseline as superiority.
Karolinska Sleepiness Scale (KSS) difference between the test and reference APAP treatments. | The patients fill KSS questionnaire immediately after each PSG study
  KSS is a simple questionnaire for subjective momentary evaluation of sleepiness/alertness [41]. A recent clinical trial [34] included subjective evaluation after polysomnography (PSG) as one of the secondary outcome measures. The KSS difference between the test treatment and baseline will not be estimated because KSS is included into the standard diagnostic PSG.
Test treatment AHI | Up to 8 weeks after study completion
  The study will test the hypothesis of the test treatment AHI being below a threshold of 9 that is within the range 5-10.

CONTACTS AND LOCATIONS:
Overall Officials: Garun Hamilton, PhD, Principal Investigator — Director of Sleep Research, Department of Respiratory & Sleep Medicine, Monash Medical Centre
Locations (1):
- Department of Respiratory & Sleep Medicine, Monash Medical Centre, Clayton, Victoria, Australia